CLINICAL TRIAL: NCT04448236
Title: Effects on Muscle Strength After Blood Flow Restriction Resistance Exercise (BFR-RE) in Early In-patient Rehabilitation of Chronic Obstructive Pulmonary Disease Acute Exacerbation (COPDAE), a Single Blinded, Randomized Controlled Study
Brief Title: Effect of Blood Flow Restriction Resistance Exercises in COPDAE In-patient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, LAU chung wai, Principal investigator, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BFR-RE in COPDAE
Record Dates: First submitted 2020-06-13; First posted 2020-06-25 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Exacerbation of COPD
Keywords: muscle strength; COPDAE; BFRRE; isometric knee extension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of the two treatment groups by drawing enclosed envelops which contain the random allocation of participants to intervention group (training with "BFR-device" and control group (training without the device). The envelopes are opened after inclusion for the individual participant only.
  Stratification of participants into two groups by maximum voluntary isometric contraction (MVIC) at baseline before randomization will be done. The cutoff for the stratification will be determined from the data in the recent service.
Who Masked: Outcomes Assessor
Masking Description: The Assessor for the primary outcome (maximum voluntary isometric contraction, MVIC) of knee extension, functional outcomes(6-minute walk test, Short Physical Performance Battery), will be blinded to the allocated study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR-RE intervention group (Experimental): The participants will have the standardised 2 week resistance training with "BFR-device" with details as follows:
  * Cuff size: medium
  * Restriction time: 5- 10 mins (stop after finishing 4 sets of training or terminating by Physiotherapists)
  * Applied location: alternate quadriceps in consecutive day
  * Applied pressure: 80% limb occlusion pressure (LOP)
  Interventions: Device: Blood flow restriction resistance exercise
- Control group (No Intervention): Same standardized 2-week in-patient rehabilitation and same amount of the above-mentioned resistance training without the "BFR device".

INTERVENTIONS:
Device: Blood flow restriction resistance exercise — Application the "Blood flow restriction device" over the proximal thigh to have 80% of the limb occlusion pressure to accumulate the metabolite generated during knee extension
  Arms: BFR-RE intervention group

SUMMARY:
This is a randomised controlled trial of the blood flow restriction resistance exercise (BFR-RE) for early rehabilitation of chronic obstructive pulmonary disease acute exacerbation (COPDAE) in the Haven of Hope Hospital.

BFR-RE was invented by Dr. Yoshiaki Sato in Japan 40 years ago. This exercise was newly introduced to the Physiotherapy Department of Haven of Hope Hospital in March, 2020 and not a routine common training in Hospital Authority. However, currently the "BFR-device" is in its 3rd generation. Under the guidance of a certified physiotherapist, a "low load intensity" can be used for resistance training to build up muscle mass and strength by applying the device over the thigh to partially limit the blood flow to the distal limb.

BFR-RE is well studied in athletes, elderlies and patients for rehabilitation after orthopaedics surgeries. A large amount of literature reveals BFR-RE with "low load intensity" shows comparable increase of muscle mass as "high load intensity" resistance training and more increase of muscle strength than those only undergoing "low load intensity" resistance training.

The objective of this study is to investigate the additional effects of 2-week BFR-RE in patients with COPDAE on top of the conventional in-patient rehabilitation training. The primary outcome is effect on localized muscle strength. The secondary outcomes include mobility function, systemic muscle strength as reflected by handgrip strength(HGS), health related quality of life, unplanned readmission to acute hospital rate within 1 month for COPDAE.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a prevalent disease around the world particularly in developed countries. COPD often has frequent admissions for acute exacerbation which increase the risks of mortality. Muscular dysfunction is one of extra-pulmonary morbidity of COPD.

Reduced muscle strength is associated with increased mortality in moderate to severe COPD. However, at least 70% of 1-repetition maximum (1-RM) of weight is needed to achieve muscle growth in resistance training. This might not be feasible particularly to the patients admitted for COPD acute exacerbation (COPDAE).

Blood flow restriction resistance training (BFR-RE), Kaatsu training, was developed by Dr. Yoshiaki Sato more than 40 years ago. The basic physiological mechanism of BFR-RE to increase muscle mass and strength is by metabolite accumulation, e.g. lactate. The metabolites lead to increase of serum growth hormone (GH) which promotes the collagen synthesis for tissue repair and recovery. The surge of GH leads to release of insulin-like growth factor (IGF-1) which is a protein related to muscle growth. IGF-1 contributes the muscle gain, which is a muscular anabolic process, by enhancing satellite cell proliferation.

Concerning growth of muscle mass, BFR-RE leads to a comparable increase when compared to high load resistance exercise (HL-RE). However, concerning increase of muscle strength, BFR-RE is less effective in gain than that in HL- RE but more effective than that in low load resistance exercise (LL-RE) alone. Therefore, BFR-RE can be considered when HL- RE is not advisable. (e.g. frail elderly, post-operative rehabilitation, etc.) BFR-RE is well studied among healthy adult, elderly and musculoskeletal rehabilitation patients, but not in COPDAE patients.

Standardized isotonic knee extension resistance training on alternate day with a load of 15-30% of 1-Repetition Maximum (1-RM) with "BFR-device" will be compared with the control arm having same set of exercise training without the device in COPDAE patient during 2-week of inpatient stay. Referred to previous study with 30% drop out rate estimation, 24 patients for each arm will be needed. Study period will be set to be 9 months or until expected recruitment achieved.

Though there no adverse risk responses were reported in published randomized controlled trials in clinical populations in the literature, there are some expected transient perceptual type responses, e.g. dizziness, limb numbness, perceived exertion, delayed onset muscle soreness. There are no significant risks of complications if BFR-RE is prescribed by certified trainers who have knowledge of appropriate protocols and contraindications to the use of occlusive stimuli.

The effect on muscle strength in COPDAE inpatient, which is not well studied in the literatures, will be the primary outcome of this study. The effect on mobility functions, systemic muscle strength, health related quality of life, unplanned readmission rate within 1 month of discharge for COPDAE, acceptability and feasibility of the BFR-RE will be evaluated as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. COPD acute exacerbation (COPDAE) as the primary diagnosis for hospitalization or transfer to pulmonary wards of the Haven of Hope Hospital
2. Able to walk under supervision
3. Understand instruction in Cantonese and can give informed consent.

Exclusion Criteria:

1. Concomitant acute cardiac event
2. Severe hypertension (BP > 180/100)
3. History of venous thromboembolism
4. History of peripheral vascular disease
5. Absence of posterior tibial or dorsalis pedal pulse
6. History of revascularization of the extremity
7. History of lymphectomies
8. Extremities with dialysis access
9. Vascular grafting
10. Current extremity infection
11. Active malignancy
12. Open fracture / soft tissue injuries
13. Amputation to the lower extremity
14. Expected hospitalization less than 2 weeks on admission
15. Medications known to increase clotting risks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: chung wai LAU, MBBS, Principal Investigator — Hospital Authority, Hong Kong
Locations (1):
- Haven of Hope Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Brandner, C. R., May, A. K., Clarkson, M. J., & Warmington, S. A. Reported Side-effects and Safety Considerations for the Use of Blood Flow Restriction During Exercise in Practice and Research. Techniques in Orthopaedics. 2018; 33(2), 114-121.
- [Background] Centner C, Wiegel P, Gollhofer A, Konig D. Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. Sports Med. 2019 Jan;49(1):95-108. doi: 10.1007/s40279-018-0994-1. PMID 30306467
- [Background] Cook SB, LaRoche DP, Villa MR, Barile H, Manini TM. Blood flow restricted resistance training in older adults at risk of mobility limitations. Exp Gerontol. 2017 Dec 1;99:138-145. doi: 10.1016/j.exger.2017.10.004. Epub 2017 Oct 5. PMID 28987643
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Manini TM, Clark BC. Blood flow restricted exercise and skeletal muscle health. Exerc Sport Sci Rev. 2009 Apr;37(2):78-85. doi: 10.1097/JES.0b013e31819c2e5c. PMID 19305199
- [Background] Sato, Y. The history and future of KAATSU Training. International Journal of KAATSU Training Research. 2005; 1(1): 1-5.
- [Background] Swallow EB, Reyes D, Hopkinson NS, Man WD, Porcher R, Cetti EJ, Moore AJ, Moxham J, Polkey MI. Quadriceps strength predicts mortality in patients with moderate to severe chronic obstructive pulmonary disease. Thorax. 2007 Feb;62(2):115-20. doi: 10.1136/thx.2006.062026. Epub 2006 Nov 7. PMID 17090575
- [Background] Van't Hul A, Harlaar J, Gosselink R, Hollander P, Postmus P, Kwakkel G. Quadriceps muscle endurance in patients with chronic obstructive pulmonary disease. Muscle Nerve. 2004 Feb;29(2):267-74. doi: 10.1002/mus.10552. PMID 14755493
- [Background] Kroemer KH, Marras WS. Towards an objective assessment of the "maximal voluntary contraction" component in routine muscle strength measurements. Eur J Appl Physiol Occup Physiol. 1980;45(1):1-9. doi: 10.1007/BF00421195. PMID 7191799
- [Background] Robles PG, Mathur S, Janaudis-Fereira T, Dolmage TE, Goldstein RS, Brooks D. Measurement of peripheral muscle strength in individuals with chronic obstructive pulmonary disease: a systematic review. J Cardiopulm Rehabil Prev. 2011 Jan-Feb;31(1):11-24. doi: 10.1097/HCR.0b013e3181ebf302. PMID 20724932
- [Background] Bernabeu-Mora R, Medina-Mirapeix F, Llamazares-Herran E, Garcia-Guillamon G, Gimenez-Gimenez LM, Sanchez-Nieto JM. The Short Physical Performance Battery is a discriminative tool for identifying patients with COPD at risk of disability. Int J Chron Obstruct Pulmon Dis. 2015 Dec 3;10:2619-26. doi: 10.2147/COPD.S94377. eCollection 2015. PMID 26664110
- [Background] Hicks RW, Denholm B. Implementing AORN recommended practices for care of patients undergoing pneumatic tourniquet-assisted procedures. AORN J. 2013 Oct;98(4):383-93; quiz 394-6. doi: 10.1016/j.aorn.2013.08.004. PMID 24075334
- [Background] Kearon C, Ageno W, Cannegieter SC, Cosmi B, Geersing GJ, Kyrle PA; Subcommittees on Control of Anticoagulation, and Predictive and Diagnostic Variables in Thrombotic Disease. Categorization of patients as having provoked or unprovoked venous thromboembolism: guidance from the SSC of ISTH. J Thromb Haemost. 2016 Jul;14(7):1480-3. doi: 10.1111/jth.13336. Epub 2016 Jun 7. No abstract available. PMID 27428935
- [Background] Jeong M, Kang HK, Song P, Park HK, Jung H, Lee SS, Koo HK. Hand grip strength in patients with chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2017 Aug 9;12:2385-2390. doi: 10.2147/COPD.S140915. eCollection 2017. PMID 28848339
- [Background] Kanada Y, Sakurai H, Sugiura Y, Arai T, Koyama S, Tanabe S. Estimation of 1RM for knee extension based on the maximal isometric muscle strength and body composition. J Phys Ther Sci. 2017 Nov;29(11):2013-2017. doi: 10.1589/jpts.29.2013. Epub 2017 Nov 24. PMID 29200647
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Takeichi N, Ishizaka S, Nishiyama M, et al. Prediction of 1 repetition maximum strength from isometric strength using Hand-Held Dynamometer for the knee extenser. Gen Rehabil, 2012; 40: 1005-1009.
- [Background] Yu R, Ong S, Cheung O, Leung J, Woo J. Reference Values of Grip Strength, Prevalence of Low Grip Strength, and Factors Affecting Grip Strength Values in Chinese Adults. J Am Med Dir Assoc. 2017 Jun 1;18(6):551.e9-551.e16. doi: 10.1016/j.jamda.2017.03.006. Epub 2017 Apr 29. PMID 28465129
- [Derived] Lau CW, Leung SY, Wah SH, Yip CW, Wong WY, Chan KS. Effect on muscle strength after blood flow restriction resistance exercise in early in-patient rehabilitation of post-chronic obstructive pulmonary disease acute exacerbation, a single blinded, randomized controlled study. Chron Respir Dis. 2023 Jan-Dec;20:14799731231211845. doi: 10.1177/14799731231211845. PMID 37976375

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Flow Restriction Resistance Exercise Intervention Group: The participants will have the standardised 2 week resistance training with "Blood flow restriction-device" with details as follows:
  * Cuff size: medium
  * Restriction time: 5- 10 mins (stop after finishing 4 sets of training or terminating by Physiotherapists)
  * Applied location: alternate quadriceps in consecutive day
  * Applied pressure: 80% limb occlusion pressure (LOP)
  Blood flow restriction resistance exercise: Application the "Blood flow restriction device" over the proximal thigh to have 80% of the limb occlusion pressure to accumulate the metabolite generated during knee extension
Period: Overall Study
Arm/Group | Blood Flow Restriction Resistance Exercise Intervention Group | Control Group
Started | 27 | 26
Completed | 20 | 25
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- BFR-RE Intervention Group: The participants will have the standardised 2 week resistance training with "BFR-device" with details as follows:
  * Cuff size: medium
  * Restriction time: 5- 10 mins (stop after finishing 4 sets of training or terminating by Physiotherapists)
  * Applied location: alternate quadriceps in consecutive day
  * Applied pressure: 80% limb occlusion pressure (LOP)
  Blood flow restriction resistance exercise: Application the "Blood flow restriction device" over the proximal thigh to have 80% of the limb occlusion pressure to accumulate the metabolite generated during knee extension
- Total: Total of all reporting groups
Arm/Group | BFR-RE Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 25 | 45
Age, Continuous [Mean (Standard Deviation); unit: year] | 74.9 (11.9) | 77.4 (8.9) | 76.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 19 | 24 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 20 | 25 | 45
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 19 (3.1) | 19.8 (3) | 19.4 (3)
Body mass index, obstruction, dyspnea, exercise (BODE) index [Median (Inter-Quartile Range); unit: units on a scale] — The BODE index scores range from 0 to 10, higher the score, higher the mortality rate at 52 months.
  The index is the sum of the scores from the 4 components:
  * Body mass index= >21 (0) ; ≤21 (+1 score)
  * Forced expiratory volume in 1 second (% of predicted to normal population)= ≥65% (0) ; 50 - 64% (+1 score) ; 36 - 49% (+2 scores); ≤35% (+3 scores)
  * Dyspnea scale: Grade 0: (0); Grade 1: (0); Grade 2: (+1 score) ;Grade 3: (+2 score); Grade 4: (+3 score)
  * Distance walked in 6 minutes ≥350 m (0); 250 - 349 m (+1 score) ; 150 - 249 m (+2 score) ; ≤149 m (+3 score)
  units on a scale | 5 [3 to 7.5] | 5 [3.5 to 7] | 5 [3 to 7.5]

OUTCOME MEASURES:

1. Primary Outcome: Change of Maximal Voluntary Isometric Contraction (MVIC) of Knee Extension of the Dominant Leg in 3 Weeks
Description: To measure the change of the force-producing capabilities of a muscle group objectively during its isometric contraction condition which means muscle group under contraction with a constant velocity of joint motion and muscle length.
  Computer dynamometer will be used to measure the MVIC of the isometric knee extension of the dominant leg.
Time Frame: baseline and 3 weeks (after 10-12 sessions of training)
Measure: Median (Inter-Quartile Range); unit: kgf
Groups:
- Blood Flow Restriction Resistance Exercise (BFR-RE) Intervention Group: The participants will have the standardised 2 week resistance training with "BFR-device" with details as follows:
  * Cuff size: medium
  * Restriction time: 5- 10 mins (stop after finishing 4 sets of training or terminating by Physiotherapists)
  * Applied location: alternate quadriceps in consecutive day
  * Applied pressure: 80% limb occlusion pressure (LOP)
  Blood flow restriction resistance exercise: Application the "Blood flow restriction device" over the proximal thigh to have 80% of the limb occlusion pressure to accumulate the metabolite generated during knee extension
Arm/Group | Blood Flow Restriction Resistance Exercise (BFR-RE) Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
kgf | 25.9 [21.3 to 30.3] | 24.7 [16.6 to 35.1]

2. Secondary Outcome: Change of Scores of Short Physical Performance Battery (SPPB) in 3 Weeks
Description: SPPB is the sum of the points from the following 3 measures, high the point, better performance
  * Time needed to walk 4m distance: less than 4.82s=4 points, 4.82-6.2s=3 points, 6.21-8.7s=2 points, >8.7s=1 point; if unable to do the walk=0 point
  * Balance test: can hold side by side stand 10s= 1 point; semi-tandem stand 10s=1 point; tandem stand 10s=2 point; tandem stand 3-9.99s=1 point; if unable to do the stand=0 point
  * Repeated chair stands test:; Participant unable to complete 5 chair stands or completes stands in >60s =0 point; If chair stand time is 16.70s or more= 1 point; If chair stand time is 13.70 to 16.69s = 2 points; If chair stand time is 11.20 to 13.69s=3 points; If chair stand time is 11.19s or less= 4 points
  Minimum score=0 Maximum score=12(best performance)
Time Frame: baseline and 3 weeks (after 10-12 sessions of training)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Blood Flow Restriction Resistance Exercise (BFR-RE) Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
score on a scale | 8.5 [6.3 to 10.8] | 7 [5 to 8.5]

3. Secondary Outcome: Change of Hand Grip Strength in 3 Weeks
Description: a non-invasive marker of systemic skeletal muscle strength and function, is assessed by handheld grip dynamometer of dominant hand
Time Frame: baseline and 3 weeks (after 10-12 sessions of training)
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Blood Flow Restriction Resistance Exercise (BFR-RE) Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
kg | 1 [0 to 2] | 2 [0 to 5.5]

4. Secondary Outcome: Change of Health Related Quality of Life in 3 Weeks
Description: Self-administered Chinese version of Chronic obstructive pulmonary disease(COPD) assessment test (CAT) It contains 8 questions and 6 points each (0 to 5). Higher score means worse health status. The Minimal clinical important difference of CAT score was 2 to 3.
  Minimum score=0 Maximum score=40 (worst health status)
Time Frame: baseline and 3 weeks (after 10-12 sessions of training)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | BFR-RE Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
units on a scale | 6.5 [0.3 to 15] | 6 [2 to 12.5]

5. Secondary Outcome: Average Pain Score of Each Training
Description: Visual analog scale (0-10) for before, immediate and 5-minute post exercise. least pain=0 ; most severe pain=10
Time Frame: pain score before, immediate and 5-minute post exercise;
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Blood Flow Restriction Resistance Exercise (BFR-RE) Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
score on a scale
  Before training | 0 [0 to 0] | 0 [0 to 0]
  Immediate after training | 3.4 [1.3 to 5.4] | 0 [0 to 0]
  5 mins after training | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Reasons of Drop-out of Blood Flow Restriction Resistance Exercise
Description: Examination the reasons of drop-out in those discontinuing the training
Time Frame: baseline to 3 weeks (after 10-12 sessions of training)
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Flow Restriction Resistance Exercise (BFR-RE) Intervention Group | Control Group
Number analyzed (Participants) | 7 | 1
Participants
  Due to contact contact precaution requirement | 3 | 0
  Due to hospitalization less than 2 weeks | 2 | 1
  Due to failure to complete training | 2 | 0

7. Secondary Outcome: Feasibility of BFR Exercise
Description: Examination of drop-out rate
Time Frame: baseline and 3 weeks (after 10-12 sessions of training)
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Flow Restriction Resistance Exercise Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
Participants | 7 | 1

8. Secondary Outcome: Unplanned Readmission Rate on 1 Month Post Discharge
Description: Unplanned readmission rate within 1 month of discharge for Chronic Obstructive Pulmonary Disease Acute Exacerbation (COPDAE)
Time Frame: 1 month after the discharge of patients in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Flow Restriction Resistance Exercise Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
Participants
  Not COPDAE related | 2 | 3
  COPDAE related | 2 | 1
  No admission | 16 | 21

9. Secondary Outcome: 6-minute Walk Test Distance Gain
Description: the distance can achieved in 6-minute walk test
Time Frame: baseline and 3 weeks (after 10-12 sessions of training)
Measure: Median (Inter-Quartile Range); unit: m
Arm/Group | Blood Flow Restriction Resistance Exercise Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
m | 5.5 [-24.5 to 55.8] | 37 [17.5 to 68.5]

10. Secondary Outcome: Acceptability of Blood Flow Restriction Resistance Exercise
Description: Measure the patient's acceptance by a 5-point categorical scale after the whole program.
  1=very dislike, 2=dislike,3=no comment, 4= like, 5=very like Lowest score=1 Highest score=5(Higher score means better acceptance)
Time Frame: Acceptance scale will be assessed immediately after the program after 3 (after 10-12 sessions of training)
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Flow Restriction Resistance Exercise Intervention Group | Control Group
Number analyzed (Participants) | 20 | 25
Participants
  Very dislike / dislike / no comment | 5 | 10
  like / very like | 15 | 15

ADVERSE EVENTS:
Time Frame: 1month
Description: acute exacerbation or hospital acquired infections
Arm/Group | BFR-RE Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/25
Other Adverse Events (participants affected / at risk) | 11/20 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BFR-RE Intervention Group (N=20) | Control Group (N=25)
COPD acute exacerbation or hospital acquired infections (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) — COPD acute exacerbation or hospital acquired infections
Others (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — accidental fall with knee injury walking limited by low back pain
insomnia (Psychiatric disorders) | 1 (1) | 0 (0) — Insomnia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT04448236/Prot_SAP_ICF_000.pdf